CLINICAL TRIAL: NCT01423656
Title: Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects by Dermal Application of a LEO 29102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LEO 29102-C06
Record Dates: First submitted 2011-07-14; First posted 2011-08-26 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 2-(6-(2-(3,5-dichloro-4-pyridyl)acetyl)-2,3-dimethoxyphenoxy)-N-propylacetamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 29102 (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 29102
  Arms: LEO 29102
Drug: Placebo — Placebo Comparator: LEO 29102 vehicle
  Arms: LEO 29102 vehicle

SUMMARY:
The principal aim of this study is to obtain safety, tolerability and pharmacokinetic data when LEO 29102 is administered cutaneously as single and multiple doses to healthy subjects.

The study is divided into one single dose part, one part to compare pharmacokinetics between gender and one multiple dose part.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be Caucasian males and females between 18 and 55 years of age and with a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
* Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations

Exclusion Criteria:

* Subjects who suffer from, or show signs of eczema or other skin lesions.
* Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity), or a marketed drug within the past 3 months prior to the first dosing occasion.
* Subjects with a significant history of drug allergy as determined by the Investigator.
* Subjects with known immunocompromised state due to treatment with immunosuppressive drugs or due to history of a disease leading to immunocompromised status.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) and change from baseline in vital signs (blood pressure, pulse rate, respiratory rate and oral body temperature), ECG, telemetry,clinical laboratory and local tolerability assessments | 7 days after last dosing

SECONDARY OUTCOMES:
LEO 29102 and metabolites in blood and urine | 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MBChB, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No